CLINICAL TRIAL: NCT00072735
Title: Improvement of Use Dependent Plasticity in Chronic Stroke Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040042; 04-N-0042
Record Dates: First submitted 2003-11-07; First posted 2003-11-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-08-15

CONDITIONS: Healthy; Cerebrovascular Accident
Keywords: Use Dependent Plasticity; Cortical Reorganization; Rehabilitation; Somatosensory Nerve; Amphetamine; Stroke; Healthy Volunteer; HV
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Procedure: Electrocardiogram

SUMMARY:
This study will examine the role of an amphetamine in improving the effect that electrical nerve stimulation has over brain flexibility associated with motor training in patients who experienced a stroke more than 1 year before. Chronic stroke is the main cause of long-term disability among adults. Previous studies have shown that electrical stimulation given over the skin may improve patients' recovery of motor function. Furthermore, it is known that amphetamines can improve the effects of sensory stimulation such as touch. Use dependent plasticity refers to a process in which the performance of simple, repetitive finger movements leads to encoding the details of those actions in the primary motor cortex of the brain. Plasticity in this sense refers to the capacity for change in the brain.

Patients 18 years of age and older who have had a stroke, who have no history of other neurological and psychiatric illnesses, and who are able to contrite and perform simple attentional tasks and other tasks may be eligible for this study. There will also be healthy participants as a control group.

Participants will have an electrocardiogram. They will also go through a practice session of about 3 hours in which they become familiar with the different tasks required in the study: motor training, pinch force, and the Jebsen-Taylor Test-which requires doing as fast as possible actions that include writing, lifting small common objects, turning pages, or lifting light or heavy objects. Then during the study, patients will be involved in a variety of sessions:

* Motor training alone for about 3 hours.
* Motor training, amphetamine (or placebo), and electrical stimulation for about 6 hours.
* Motor training, amphetamine, and no electrical stimulation for about 6 hours.

A magnetic resonance imagining (MRI) scan will be done. Patients will lie still on a table that can slide in and out of a metal cylinder surrounded by a strong magnetic field. Scanning time varies from 20 minutes to 3 hours, with most scans lasting between 45 and 90 minutes. Patients may be asked to lie still for up to 60 minutes at a time. As the scanner takes pictures, there will be loud knocking noises, and the patients will wear earplugs to muffle the sound. Patients will be able to communicate with the MRI staff at all times during the scan and may ask to be moved out of the machine at any time.

During another procedure called transcranial magnetic stimulation (TMS), a wire coil will be held over the scalp. A brief electrical current will be passed through the coil, creating a magnetic pulse that stimulates the brain. Patients will hear a click and may feel a pulling sensation on the skin under the coil. There may be muscle twitches of the face, arm, or leg. Patients may be asked to tense certain muscles slightly or perform other simple actions so that the coil can be positioned appropriately. The stimulation is usually not painful, although sometimes strong contractions of the scalp muscles can cause discomfort or a headache. Patients can ask to have the procedure discontinued at any time.

For the electrical stimulation procedure, three pairs of electrodes will be placed on the skin. A quite brief pulse of current will pass between the electrodes, creating the electrical field that activates the brain. Patients will feel a brief stinging around the electrodes. Regarding the amphetamine, patients will take it orally on up to four different occasions. Usually they will take 10 mg of Dexedrin before testing.

DETAILED DESCRIPTION:
OBJECTIVES:

There is no universally accepted strategy to promote recovery of motor function after chronic stroke, the main cause of long-term disability among adults. It is desirable to develop strategies to enhance motor training in this patient group. A recent study in stroke patients and healthy volunteers demonstrated that somatosensory nerve stimulation prior to motor training leads to improvements in use-dependent plasticity (UDP), a process thought to underlie recovery of motor function after brain injury (Sawaki et al., unpublished information). Interestingly, the effects of sensory input on cortical plasticity can be enhanced by a single dose of amphetamine. The objective of this protocol is to further enhance the effect that somatosensory nerve stimulation has on motor training by means of pre-medication with amphetamine. This effect over motor training will be measured by the magnitude of training-induced UDP. Our hypothesis is that the amphetamine-enhanced effects of somatosensory nerve stimulation will increase the magnitude of training-induced UDP.

STUDY POPULATION:

We plan to study 24 patients with chronic strokes and 24 healthy age- and gender matched normal volunteers.

DESIGN:

All subjects will participate in 5 different randomized sessions on separate days. The first session will be a familiarization with the behavioral tasks. A second experiment will consist of training with no further interventions to obtain baseline UDP changes. In another two sessions, subjects will be premedicated in a blind manner with amphetamine or placebo before administration of somatosensory nerve stimulation followed by motor training to induce UDP. In the last experiment, the participants will be premedicated with amphetamine and will be exposed to sham somatosensory stimulation prior to the motor training to induce UDP.

OUTCOME MEASURES:

Primary outcome measure will be the magnitude of UDP (training-induced changes in transcranial magnetic stimulation-evoked kinematic responses). Secondary outcome measures are pinch force; and a functional measure of activities of daily life (ADL): Jebsen-Tailor-Test. To better understand the mechanisms underlying the proposed behavioral gains, we will use TMS to identify changes in corticomotor excitability.

ELIGIBILITY:
* INCLUSION CRITERIA:

We will include patients with thromboembolic non-hemorrhagic hemispheric lesions at least 12 months after the stroke.

We will choose patients who initially had a severe motor paresis (below MRC grade 2), which subsequently recovered to the point that they have a residual motor deficit but can perform the required tasks.

As a control group, we will include age- and gender matched normal volunteers with matched non-dominant/dominant hand (to the affected hand of the stroke patients).

EXCLUSION CRITERIA:

Patients with more than one stroke in the middle cerebral artery territory.

Patients with bilateral motor impairment.

Patients with cerebellar or brainstem lesions.

Patients receiving alpha-adrenergic antagonists or agonists, major/minor tranquilizers, clonidine, prazosin, phonation, benzodiazepines, scopolamine, haloperidol, other neuroleptics, barbiturates and MAO inhibitors.

Patients or normal volunteers unable to perform the task (wrist or elbow flexion at least MRC grade 2).

Patients or normal volunteers with history of severe alcohol or drug abuse, psychiatric illness like severe depression, poor motivational capacity, or severe language disturbances, particularly of receptive nature or with serious cognitive deficits (defined as equivalent to a mini-mental state exam score of 23 or less).

Patients or normal volunteers with severe uncontrolled medical problems (e.g. hypertension, cardiovascular disease, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, or a deteriorated condition due to age, uncontrolled epilepsy or others).

Patients or normal volunteers with increased intracranial pressure as evaluated by clinical means.

Patients or normal volunteers with unstable cardiac arrhythmia.

Patients or normal volunteers with history of hyperthyroidism or individuals receiving drugs acting primarily on the central nervous system.

Patients and normal volunteers with more than moderate to severe microangiopathy, polyneuropathy, diabetes mellitus, or ischemic peripheral disease.

Pregnancy.

Patients and normal volunteers less than 18 years of age.

Lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2003-11-06; Study Completion 2007-08-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Conforto AB, Kaelin-Lang A, Cohen LG. Increase in hand muscle strength of stroke patients after somatosensory stimulation. Ann Neurol. 2002 Jan;51(1):122-5. doi: 10.1002/ana.10070. PMID 11782992